CLINICAL TRIAL: NCT03463096
Title: Advanced Gravitational Physiology the Lung Under High-G Acceleration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Oxford (Other); QinetiQ Ltd (Industry); UK Space Agency (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SP801
Record Dates: First submitted 2018-02-28; First posted 2018-03-13 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-02

CONDITIONS: Respiratory Physiology
Keywords: respiratory; physiology; gravity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Centrifuge study (Experimental): High G acceleration on a long-arm human centrifuge
  Interventions: Other: High G acceleration on a long-arm human centrifuge

INTERVENTIONS:
Other: High G acceleration on a long-arm human centrifuge — Gx (chest-to-back) and Gz (head-to-toe)

SUMMARY:
This is a study of advanced lung physiology in altered gravitational conditions, consisting of respiratory measurements in healthy volunteers during high G acceleration on a long-arm human centrifuge.

DETAILED DESCRIPTION:
The lung is highly gravity-dependent - it has little actual tissue mass and deforms under its own weight. This is relevant to astronauts in space, but is actually much more broadly important to life on Earth. Every time we change our posture - for example from lying to standing - the direction in which gravity acts across the lung changes. These postural effects can become clinically important in critically ill patients. Currently there is debate in the scientific world about how gravity actually influences lung function, and how it interacts with other factors such as the anatomical structure of the airways and blood vessels of the lung. New technology developed by researchers at the University of Oxford now has the potential to help answer some of these questions. This device uses a technique called laser absorption spectroscopy to make measurements of breathing gases that are much more accurate than previous techniques - it is able to count the number of oxygen, carbon dioxide and water vapour molecules in and out while a person breathes. A non-invasive 15-minute breathing test with this technology provides information on the distributions of airflow and blood flow in the lungs, and it has been deployed successfully in the operating theatre and in intensive care units. This study aims to make comprehensive measurements of lung physiology under altered gravitational conditions and develop the technology and measurement techniques for possible future use in microgravity. This will include measurements of oxygen and carbon dioxide from the laser gas analyser (and measures of lung inhomogeneity obtained from these), lung mechanics and breathing drive.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer who has provided informed consent

Exclusion Criteria:

* any significant medical problem, as documented extensively in the study ethics documentation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Lung inhomogeneity index | Determined over a 15-minute multi-breath washout at 3 G on the centrifuge
  The lung inhomogeneity index is the standard deviation for the natural logarithm of the standardised lung compliance, equivalent to the standard deviation for the natural logarithm of the ratio between fractional lung compliance and fractional alveolar volume of the lung units.
  It is determined using the respiratory data obtained by molecular flow sensing using the laser gas analyser.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Smith, Principal Investigator — King's College London
Locations (1):
- Centre of Human and Aerospace Physiological Sciences, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No